CLINICAL TRIAL: NCT01032954
Title: Phase Iv Study On The Safety And Efficacy Of The Full Face Applications Of Variable Doses Of 125 To 250 Units Of A Commercial Botulinum Toxin Type A (Dysport®)
Brief Title: Safety and Efficacy of the Full Face Applications of Variable Doses of a Commercial Botulinum Toxin Type a (Dysport®)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hexsel Dermatology Clinic (Other)
Responsible Party: Principal Investigator, Doris Hexsel, MD, Hexsel Dermatology Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-CBED09-02
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Results first posted 2020-09-17 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Sun-induced Wrinkles
Keywords: Botulinum Toxin; Rejuvenation; Facial dynamic wrinkles
MeSH Terms: interventions — Botulinum Toxins; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 125 to 170 IU of "'Botulinum toxin' " (Active Comparator): group with intervention of 125 to 170 IU of 'Botulinum toxin'
  Interventions: Drug: Botulinum toxin
- 171 to 210 IU of 'Botulinum toxin' (Active Comparator): Patients who have received 171 to 210 IU of 'Botulinum toxin'
  Interventions: Drug: Botulinum toxin
- 211 to 250 IU of Botulinum toxin (Active Comparator): Patients who have received 211 to 250 U of Botulinum toxi'
  Interventions: Drug: Botulinum toxin

INTERVENTIONS:
Drug: Botulinum toxin — Drug: Botulinum toxin
  Indications for eligibility and total doses that will be applied in each part of the face, at visit 1:
  Upper face:
  * Crow's feet wrinkles - 70 units
  * Glabella - 50 units
  * Forehead - 40 units
  Mid face:
  * Lower eyelid - 5 units
  * Nasal wrinkles - 20 units
  * Malar wrinkles - 10 units
  Lower face:
  * Peri-oral wrinkles - 15 units
  * Asymmetric smile or gummy smile - 5 units
  * "Cellulitic chin" - 20 units
  * Marionette lines - 25 U According to the patients needs, the doses can vary ±10% in terms of the amount of units that will be injected.
  Patients will be allocated in each group and receive the doses described above at visit 1. At visit 2, all the patients will receive a touch-up of a standard dose of 25 U, distributed on the treated areas according patient's needs.
  Other Names: Dysport

SUMMARY:
This is an open-label and phase IV study of full face injections of variable doses of botulinum toxin type A (BT-A). As it is an open-label and not blind study, both investigator and subjects will know the injection local and doses of the study drug. Patients will be randomized into 3 different groups. Each group will receive a specific dose according with the indication evaluated by the investigator. Six visits will be schedule in this study.

DETAILED DESCRIPTION:
4.2 Methodology

4.2.1 Patient evaluation After providing written informed consent, subject's eligibility will be assessed at a Screening Visit. The subject's general medical history will be recorded. This includes demographic data, history of surgical and cosmetic procedures, dermatological assessment, physical examination, and prior concomitant medications. A pregnancy test will also be performed.

4.2.1.1 Severity of wrinkles

One sub-investigator will rate the wrinkles with the following validated severity scales for the main areas of the face at Baseline, Week 4, Week 8, Week 16 and Week 24:

* Clinical 0-3 score for standardized assessment of facial wrinkles in the glabella area (from GLADYS study)
* Photometric Atlas for the Assessment of Crow's Feet Severity
* Facial Wrinkle Scale, for forehead lines (Carruthers A, et al. Dermatol Surg. 2003;29(5):461-7)

4.2.1.2 Standard set of photographs will be taken

At Screening , 2, 3, 4 and 5 visits, photographs will be taken:

All the photographs will be taken in a standardized photographic mode with fixed position of the camera. A guideline with examples of standardized photos with delimit standardized positions will be provided to the person responsible to take the photos.

In the photographs, each research subject will be identified by a tag containing a reference to the study, the number of the research subject and the control date. The research subjects should wash their faces before the photographic procedure to remove excess oil and all make up will be removed. All the pictures will be taken at the same room and under same parameters.

The photograph set consist of

* Full face frontal view relaxed;
* One set of photographs relaxed and contracted of each indication that patient will be or was treated in this study.

At the end of the study, two independent evaluators (dermatologists) will assess before and after pictures in a blinded manner. This evaluation will be done to assess the efficacy of BT-A in the injected areas not assessed by the scales.

4.2.3 Groups of treatment

Subjects will be assigned to one of the three following treatment groups, according with the total dose received in visit 1:

* Group 1: 30 subjects who received 125 to 170 U of BT-A (Dysport®)
* Group 2: 30 subjects who received 171 to 210 U of BT-A (Dysport®)
* Group 3: 30 subjects who received 211 to 250 U of BT-A (Dysport®)

4.2.4 Reconstitution of the study product and Treatment Administration An independent, experienced and registered pharmacist will be the assigned to carry through the reconstitution of the products. She will prepare the dilutions and the syringes of the product (DYSPORT®) immediately prior to the injections.

The dilutions of DYSPORT® 500 units per vial will be made with 2 mL of 0.9% sterile saline, using 3 mL syringes and a 21 gauge needle, giving a concentration of 250 units/mL or 2.5 units/0.01 mL of the reconstituted product.

An experienced dermatologist in the use of botulinum toxins (principal investigator - DH) will perform all the injections according to the indications and total number of units that will be injected according to the treatment plan, which aims to obtain the best results. She will only perform the injections and will not participate in other phases of this study.

The application of the BT-A will be made with Becton, Dickinson and Company (BD) Ultra-fine II 0.3 cc syringes, with a 29 gauge needle, 0.5 cm in length (short needle).

Immediately after the application, the side effects will be verified and if needed, will be registered and managed.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent;
2. Subjects aged between 30 and 60 years;
3. Skin Fitzpatrick Phototypes I to VI;
4. Subjects that never received BT-A or who had previous injections of BT-A in no more than one third of the face with in the last 6 months;
5. Subjects presenting at least two indications for treatment with BT-A in each third of the face;
6. Medical history and physical examination which, based on the investigator's opinion, do not prevent the patient from taking part in the study and use the product under investigation;
7. Subjects of childbearing age should present a negative urine pregnancy test (instant test) at baseline and should be using an effective contraceptive method (oral or injectable contraceptive, for at last three months, and use of preservative; subjects with: hysterectomy, oophorectomy or tubal ligation);
8. Availability of the patient throughout the duration of the study (24 weeks);
9. Subjects that agree not to undergo other cosmetic or dermatological procedures during the study;
10. Subjects with sufficient schooling and awareness to enable them to cooperate to the degree required by the study protocol.

Exclusion Criteria:

1. Pregnant women or women intending to become pregnant during the study;
2. Subjects participating in other clinical trials;
3. Presence of scars on the face that may interfere with the result of study;
4. Subjects with neoplastic, muscular or neurological diseases;
5. Concurrent use of treatments that affect neuromuscular transmission, such as curare-like depolarizing agents, lincosamides, polymyxins, anticholinesterases affecting the striated muscle and aminoglycoside antibiotics.
6. Subjects with inflammation or active infection in the face;
7. Subjects with a history of sensitivity to the components of the formula;
8. Subjects with prior history of eyelid ptosis; marked facial asymmetry, excessive dermatochalasis, deep dermal scarring or thick sebaceous skin.
9. Subjects presenting myasthenia gravis, Eaton-Lambert Syndrome and motor neuron diseases;
10. Subjects with coagulation disorders or using anticoagulants;
11. Subjects with known systemic autoimmune diseases;
12. Subjects clinically diagnosed anxiety disorder or any significant psychiatric disorder (e.g. depression) that, in the opinion of the Evaluator, might interfere with the Subject's participation in the study;
13. Subjects with a history of medical treatment non-adherence or showing unwillingness to adhere to the study protocol.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris M Hexsel, MD, Principal Investigator — Brazilian Center for Studies in Dermatology
Locations (1):
- Brazilian Center for Studies in Dermatology, Porto Alegre, Rio Grande do Sul, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- 125 to 170 Units of Botulinum Toxin Type A: Subjects have received the lower dose of Botulinum Toxin type A
- 171 to 210 Units of Botulinum Toxin Type A: Subjects have received the intermediate dose of Botulinum Toxin type A.
- 211 to 250 Units of Botulinum Toxin Type A: Subjects have received the higher dose of Botulinum Toxin type A.
Period: Overall Study
Arm/Group | 125 to 170 Units of Botulinum Toxin Type A | 171 to 210 Units of Botulinum Toxin Type A | 211 to 250 Units of Botulinum Toxin Type A
Started | 30 | 30 | 30
Completed | 26 | 29 | 30
Not Completed | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Subjects have received the lower dose of Botulinum Toxin type A, between 125 to 170 units of Botulinum Toxin type A.
- Group 2: Subjects have received the intermediate dose of Botulinum Toxin type A, between 171 to 210 units of Botulinum Toxin type A.
- Group 3: Subjects have received the higher dose of Botulinum Toxin type A, between 211 to 250 units of Botulinum Toxin type A
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 30 | 30 | 30 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 30 | 90
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (9) | 47 (9) | 50 (9) | 48 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 30 | 90
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 30 | 30 | 30 | 90

OUTCOME MEASURES:

1. Primary Outcome: Wrinkles' Severity (Forehead)
Description: Facial Wrinkle Scale: 0 - none, 1 - mild; 2 - moderate; 3 - severe
Time Frame: Baseline; Week 4; Week 16; Week 20; Week 24
Population: Patients in each visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- 125 to 170 Units of Botulinum Toxin Type A: Subjects were treated with a total dose of 125 to 170 units of Botulinum Toxin type A on facial indications in upper, middle and lower face.
- 171 to 210 Units of Botulinum Toxin Type A: Subjects were treated with a total dose of 171 to 210 units of Botulinum Toxin type A on facial indications in upper, middle and lower face.
- 211 to 250 Units of Botulinum Toxin Type A: Subjects were treated with a total dose of 211 to 250 units of Botulinum Toxin type A on facial indications in upper, middle and lower face.
Arm/Group | 125 to 170 Units of Botulinum Toxin Type A | 171 to 210 Units of Botulinum Toxin Type A | 211 to 250 Units of Botulinum Toxin Type A
Number analyzed (Participants) | 26 | 29 | 30
units on a scale
  Baseline | 2.31 (0.84) | 2.66 (0.49) | 2.60 (0.68)
  Week 4 | 1.78 (0.44) | 1.33 (0.70) | 0.93 (0.70)
  Week 16 | 1.82 (0.75) | 2.15 (0.75) | 1.96 (0.66)
  Week 20 | 2.25 (0.89) | 2.48 (0.68) | 2.32 (0.61)
  Week 24 | 2.44 (0.88) | 2.58 (0.58) | 2.48 (0.63)
Statistical Analysis 1: Comparison: 125 to 170 Units of Botulinum Toxin Type A vs 171 to 210 Units of Botulinum Toxin Type A vs 211 to 250 Units of Botulinum Toxin Type A; Test type: Superiority or Other; p < 0.05, GLM= GENERAL LINEAR MODELS WITH REPEATED — P-value threshold for significance: <0.05

2. Primary Outcome: Wrinkles' Severity (Glabella)
Description: GLADYS study Atlas: 0 - no wrinkles, 1 - mild wrinkles; 2 - moderate wrinkles; 3 - severe wrinkles
Time Frame: Baseline; Week 4; Week 16; Week 20; Week 24
Population: Patients in each visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 125 to 170 Units of Botulinum Toxin Type A | 171 to 210 Units of Botulinum Toxin Type A | 211 to 250 Units of Botulinum Toxin Type A
Number analyzed (Participants) | 26 | 29 | 30
units on a scale
  Baseline | 1.92 (0.67) | 2.07 (0.53) | 2.20 (0.66)
  Week 4 | 0.54 (0.58) | 0.59 (0.50) | 0.57 (0.50)
  Week 16 | 1.25 (0.60) | 1.12 (0.60) | 1.07 (0.54)
  Week 20 | 1.42 (0.65) | 1.44 (0.58) | 1.31 (0.71)
  Week 24 | 1.65 (0.69) | 1.66 (0.48) | 1.53 (0.63)
Statistical Analysis 1: Comparison: 125 to 170 Units of Botulinum Toxin Type A vs 171 to 210 Units of Botulinum Toxin Type A vs 211 to 250 Units of Botulinum Toxin Type A; Test type: Superiority or Other; p < 0.05, GLM — P-value threshold for significance: <0.05

3. Primary Outcome: Wrinkles' Severity (Periocular [Crow's Feet])
Description: Photonumeric Atlas for the Assessment of Crow's Feet Severity: 0 - none, 1 - mild; 2 - moderate; 3 - severe
Time Frame: Baseline; Week 4; Week 16; Week 20; Week 24
Population: Patients in each visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 125 to 170 Units of Botulinum Toxin Type A | 171 to 210 Units of Botulinum Toxin Type A | 211 to 250 Units of Botulinum Toxin Type A
Number analyzed (Participants) | 26 | 29 | 30
units on a scale
  Baseline | 2.04 (0.72) | 2.41 (0.57) | 2.17 (0.79)
  Week 4 | 1.04 (0.66) | 1.21 (0.56) | 1.27 (0.45)
  Week 16 | 1.54 (0.59) | 1.92 (0.49) | 1.86 (0.71)
  Week 20 | 1.67 (0.70) | 2.12 (0.44) | 2.10 (0.41)
  Week 24 | 1.88 (0.59) | 2.10 (0.41) | 2.33 (0.55)

ADVERSE EVENTS:
Arm/Group | 125 to 170 Units of Botulinum Toxin Type A | 171 to 210 Units of Botulinum Toxin Type A | 211 to 250 Units of Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/26 | 0/29 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No